CLINICAL TRIAL: NCT02708927
Title: Emotional Processing, Family Life, Friendship and Social Integration in Patients With Multiple Sclerosis
Acronym: EMOSOCIAL-MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: FONDATION POUR L'AIDE A LA RECHERCHE SUR LA SCLEROSE EN PLAQUES (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2015/11
Record Dates: First submitted 2016-03-10; First posted 2016-03-15 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Multiple Sclerosis
Keywords: social integration; cognitive impairment; emotional processing; quality of life
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patient (Experimental): MS diagnosis according to McDonald criteria (Polman et al., 2005). Relapsing-remitting MS (RRMS) according to Lublin et al. (1996);
  Interventions: Other: Clinical evaluation; Other: Cognitive evaluation
- Control (Experimental): healthy subject
  Interventions: Other: Cognitive evaluation

INTERVENTIONS:
Other: Clinical evaluation — • Clinical assessment : Expanded Disability Status Scale (EDSS), ambulation test. Medications will be recorded.
  Arms: patient
Other: Cognitive evaluation — • Neuropsychological, psychological, social and social cognitive evaluation

SUMMARY:
In addition to the physical, cognitive and psychological symptoms experienced by individuals with Multiple Sclerosis (MS), there is new research which indicates that some individuals with MS have a deficit in emotional processing, specifically, facial affect recognition. Emotional processing is defined as "a central aspect of social cognition". Models of social cognition indicate that emotional processing is an essential component of interpersonal relationships. The failure to accurately perceive other's emotions has been shown to lead to difficulty in social relationships, misinterpreting other's affect, and consequently, inappropriate responding.

However, even though a significant number of individuals with MS have impairments in emotional processing, we do not yet have an understanding of how these impairments affect the social functioning of individuals with MS, including the impact of these deficits on family structure. It is well-known that MS impacts one's social functioning including factors such as employment, daily living activities and interpersonal relationships. Recently a strong correlation was observed between reduced social participation in MS and quality of life. There is evidence to suggest that emotional processing deficits lie at the heart of this reduced social participation in persons with MS, leading to decreased social functioning and thus reduced quality of life. However, to date, this hypothesis has not been tested.

ELIGIBILITY:
Inclusion Criteria (patient group):

* Age 18-45 years;
* MS diagnosis according to McDonald criteria (Polman et al., 2005);
* RRMS;
* Disease duration < 15 years;
* Fluent French speaker;
* Have a significant other (family members or close friends) who was willing to complete the informant questionnaire BAFQ;
* Being affiliated to health insurance;
* Having signed an informed consent (later than the day of inclusion and before any examination required by research).

Inclusion Criteria (healthy control):

* Age 18-45 years
* Fluent French speaker;
* Have a significant other (family members or close friends) who was willing to complete the informant questionnaire BAFQ.
* Being affiliated to health insurance
* Having signed an informed consent (later than the day of inclusion and before any examination required by research)

Exclusion Criteria (patient group):

* Other progressive neurological disease;
* psychiatric comorbidity including severe depression according to Diagnostic and Statistical Manual-IV (DSM-IV);
* alcohol or other addiction to toxic;
* EDSS> 6;
* Disabling visual or motor problems preventing participation to neuropsychological assessments;
* relapse since less than one month;
* change of disease-modifying therapy or psychotropic drug since less than three month;
* change of psychotropic drug since less than one month;
* Prior neuropsychological testing with the same tests less than one year prevents the participant to participate at this study.
* Illiteracy, is unable to count or to read;
* Being under guardianship.
* Pregnant or breastfeeding women;

Exclusion Criteria (healthy control):

* History of neurological disease;
* family history of MS;
* psychiatric comorbidity including severe depression according to DSMIV;
* alcohol or other toxic addiction;
* usage of psychotropic drugs;
* Known cognitive complaint or neuropsychological affection;
* Prior neuropsychological testing with the same tests less than one year prevents the participant to participate at this study.
* Illiteracy, is unable to count or to read;
* Being under guardianship.
* Pregnant or breastfeeding women;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2016-03-03 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Interaction between measures of emotional processing (z score) and functional measures of social interaction | At inclusion (day 0)
  among the 3 groups (impaired MS, no impaired MS and HS)

SECONDARY OUTCOMES:
Correlation between measures of emotional processing with cognitive testing (z scores by domain) and cognitive functioning evaluated by significant other | At inclusion (day 0)
  (BAFQ)
Correlation between measures of emotional processing and quality of life measures | At inclusion (day 0)
  (MUSIQoL questionnaire).
Impact of the cognitive impairment on the relationship of emotional processing (z score) with interpersonal relationships (family, friendship, marital) and society integration and social functioning. | At inclusion (day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno BROCHET, Prof, Principal Investigator — University Hospital, Bordeaux
Locations (2):
- France (2):
  - CHU de Bordeaux, Bordeaux
  - CHU de Dijon, Dijon